CLINICAL TRIAL: NCT06545994
Title: A Prospective Cohort Study on the Dynamic Monitoring of Serum Kisspeptin Levels Throughout Pregnancy and Exploring Its Predictive Value for Gestational Diabetes Mellitus in PCOS Patients
Brief Title: A Prospective Cohort Study on the Serum Kisspeptin Levels Throughout Pregnancy in PCOS
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhang Wei, Professor, Ph.D, Fudan University
Other Study IDs: FudanU2024-04-07
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Polycystic Ovary Syndrome; Pregnancy Complications
Keywords: Polycystic Ovary Syndrome; Pregnancy Complications; Kisspeptin; gestational diabetes mellitus; insulin resistance
MeSH Terms: conditions — Polycystic Ovary Syndrome; Pregnancy Complications; Diabetes, Gestational; Insulin Resistance | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum kisspeptin, insulin, testosterone and blood glucose in the first trimester, second trimester and late pregnancy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCOS group: Pregnant women between 18 and 40 years old who were diagnosed as polycystic ovary syndrome before pregnancy, registered in the OB & GYN Hospital of Fudan University for prenatal check during the first trimester. The diagnostic criteria for PCOS are based on the 2003 Rotterdam diagnostic criteria.
  Exclude healthy women with all other diseases that may have ovulation disorders or hyperandrogenism; There are other serious illnesses or complications present; Other endocrine disorders exist: thyroid diseases such as hyperthyroidism or hypothyroidism; During pregnancy, medication that may affect Kisspeptin or insulin levels, such as metformin or insulin therapy, is being used;
  Interventions: Other: Observation
- Control group: Healthy pregnant women between 18 and 40 years old women without a history of PCOS.
  Exclude healthy women with all other diseases that may have ovulation disorders or hyperandrogenism; There are other serious illnesses or complications present; Other endocrine disorders exist: thyroid diseases such as hyperthyroidism or hypothyroidism; During pregnancy, medication that may affect Kisspeptin or insulin levels, such as metformin or insulin therapy, is being used;

INTERVENTIONS:
Other: Observation — It's a observational cohort study and no interventions are performed.
  Groups: PCOS group

SUMMARY:
The current study aims to investigate the dynamic serum kisspeptin levels throughout pregnancy and to explore its predictive value for GDM in PCOS.

DETAILED DESCRIPTION:
The current prospective cohort study aims to investigate the dynamic serum kisspeptin levels in the patients with polycystic ovary syndrome (PCOS) at different trimesters of pregnancy, to analyze the associations between serum kisspeptin, insulin, glucose and testosterone, and to explore the predictive value of kisspeptin for GDM and other complications in PCOS patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years old
* Women diagnosed as PCOS who register for prenatal check ups in the obstetrics outpatient department of hospitals during early pregnancy.(The diagnostic criteria for PCOS are based on the 2003 Rotterdam diagnostic criteria (any two out of the three key characteristics of PCOS: oligo-amenorrhea, hyperandrogenism, and polycystic-appearing ovarian morphology on ultrasonography) .

Exclusion Criteria:

* All other diseases with ovulation disorders or hyperandrogenism

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Positive pregnancy test and confirmed intrauterine singleton pregnancy by ultrasound
Study Population: The characteristics of patients with polycystic ovary syndrome include amenorrhea or infrequent menstruation, high hormone levels, and polycystic ovary like changes in the ovaries. Usually accompanied by fertility disorders and metabolic disorders, PCOS patients face a higher risk of pregnancy complications during pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Dynamic changes of serum kisspeptin levels throughout pregnancy in PCOS patients | 40 weeks
  Serum kisspeptin levels in the first, second trimester and late pregnancy of PCOS patients and control group.

SECONDARY OUTCOMES:
The association between serum Kisspeptin levels and the prevalence of GDM in PCOS patients | 40 weeks
  The predictive value of serum Kisspeptin levels in the first trimester for GDM in PCOS patients
The association between serum Kisspeptin levels and the prevalence of insulin resistance in PCOS patients | 40 weeks
  The predictive value of serum Kisspeptin levels in the first trimester for insulin resistance in PCOS patients

CONTACTS AND LOCATIONS:
Overall Officials: Hexia Xia, M.D., Principal Investigator — The Obstetrics & Gynecology Hospital of Fudan University
Locations (1):
- OB & GYN Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided